CLINICAL TRIAL: NCT01070680
Title: Dexmedetomidine vs Placebo in ERCP Sedation.A Randomized Pilot Study
Brief Title: Dexmedetomidine Versus Placebo in Endoscopic Retrograde Cholangiopancreatography (ERCP) Sedation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Maxim Mazanikov, MD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: a004c; 2009-014862-25 (EudraCT Number)
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Pancreatitis
Keywords: ERCP; dexmedetomidine; propofol; patient-controlled sedation; Chronic Alcoholic pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine (Active Comparator): sedative medicine
  Interventions: Drug: Precedex
- sodium chloride 0,9% (Placebo Comparator)
  Interventions: Drug: sodium chlorid 0,9%

INTERVENTIONS:
Drug: Precedex — mkg/ml,continuous infusion at rate 0.7 µg/kg/h
  Other Names: dexmedetomidine hydrochloride injection
  Arms: dexmedetomidine
Drug: sodium chlorid 0,9% — continuous intravenous infusion
  Other Names: NaCl 0,9%
  Arms: sodium chloride 0,9%

SUMMARY:
In this pilot prospective non-commercial clinical trial the investigators will study the use of dexmedetomidine as an adjuvant to the patient-controlled propofol sedation in a placebo-controlled and randomized manner in patients with drug addiction during Endoscopic Retrograde Cholangiopancreatography (ERCP). Dexmedetomidine is a sedative medication used mostly in intensive care units,and is marketed under the brand name Precedex. Dexmedetomidine has sedative, analgesic, sympatholytic, and anxiolytic properties. It produces sedation without causing significant respiratory depression. Recent research has suggested dexmedetomidine to be effective in treatment of alcohol withdrawal signs. In previous studies dexmedetomidine was insufficient as an only sedative agent in ERCP and colonoscopy, but it has not been assessed for sedation in patients with chronic pancreatitis. The main objective of this trial is to evaluate if dexmedetomidine can reduce propofol and opioid consumption and facilitate the performance of ERCP in patients with chronic pancreatitis due to drug addiction.Secondary objectives of the trial are the stability of vital signs and safety, patients´ satisfaction plus recovery time from sedation.

50 elective ERCP patients with chronic pancreatitis after written informed consent and randomisation will be recruited to the study. Exclusion criteria are:allergy to propofol, opioid or dexmedetomidine, ASA class greater than 3. All the patients will receive patient-controlled propofol sedation. In dexmedetomidine group dexmedetomidine infusion will be started before sedation beginning and in placebo group placebo-solution (NaCl0,9%) will be administered in the similar manner.Standard monitoring for vital signs will be applied,also sedation degrees will be evaluated with sedation scores. At the end of procedure total amount of propofol and opioid will be calculated,patients and endoscopists satisfaction and the difficulty of ERCP will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Elective ERCP-patients with chronic alcohol pancreatitis

Exclusion Criteria:

* Allergy to the dexmedetomidine, propofol or any opioid, ASA(American Society of Anaesthesiology)class grater when 3

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
sedation degree | 1 day
propofol consumption | 1 day
endoscopist´s and patient´s satisfaction | 1 day
vital signs:blood pressure, oxygen saturation, heart rate, breathing rate | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Maxim Mazanikov, MD, Principal Investigator — Helsinki University Central Hospital,Department of Anaesthesiology; Marianne Udd, MD,PhD, Principal Investigator — Helsinki University Central Hospital,Department of Surgery; Outi Lindström, MD, Principal Investigator — Helsinki University Central Hospital,Department of Surgery; Leena Kylänpää, Docent, Principal Investigator — Helsinki University Central Hospital,Department of Surgery; Jorma Halttunen, Docent, Principal Investigator — Helsinki University Central Hospital,Department of Surgery; Martti Färkkilä, Professor, Principal Investigator — Helsinki University Central Hospital,Department of Gastroenterology; Reino Pöyhiä, Docent, Study Director — Helsinki University Central Hospital,Department of Anaesthesiology; Harri Mustonen, PhD, Principal Investigator — Department of Gastrointestinal and General Surgery, Helsinki
Locations (1):
- Helsinki University Central Hospital,Meilahti hospital,Endoscopy unit, Helsinki, Uusimaa, Finland